CLINICAL TRIAL: NCT00967421
Title: Development of a Valid Test Battery for Assessing Driving Ability When Influenced by Drugs.
Acronym: VALIDAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: SINTEF Health Research (Other); Norwegian University of Science and Technology (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ES437291 VALIDAD
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Automobile Driving
Keywords: Driving; DUI; Driving simulation; Drugs; Ethanol
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAC 0.5 (Experimental): BAC level 0.5 g/dL (drink + placebo pill)
  Interventions: Drug: ethanol
- BAC 1.0 (Experimental): BAC level 1.0 g/dL (drink + placebo pill)
  Interventions: Drug: Ethanol
- placebo (Placebo Comparator): BAC level 0,0 g/dL (placebo drink+ placebo pill)
  Interventions: Other: Placebo drink

INTERVENTIONS:
Drug: ethanol — BAC level 0.5 g/dL (drink + placebo pill). Drink with 2,4 grams per kilo body weight, administered orally during 60 min, administration ending 30 min prior to start of testing. Placebo pill.
  Arms: BAC 0.5
Drug: Ethanol — BAC level 1.0 g/dL (drink + placebo pill). Drink with 3,6 grams per kilo body weight, administered orally during 60 min, administration ending 30 min prior to start of testing. Placebo pill.
  Arms: BAC 1.0
Other: Placebo drink — Placebo drink containing no alcohol + placebo pill
  Arms: placebo

SUMMARY:
The purpose of the validation study is to develop a valid test battery for assessing driving ability in a driving simulator when influenced by drugs. Ethanol has known, well-documented and well-characterized effects on driving behaviour and accident risk, and will be used to assess the simulator test scenarios' sensitivity to drug effects. Once the test scenarios have been refined and their ability to predict driving accident risk have been validated, we plan to use the simulator to assess driving ability under the influence of different drugs suspected to produce driving impairment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, caucasian males aged 25-50 years in possession of a valid driver's license for the last 5 years.
* Recreational alcohol drinkers without alcohol dependence or abuse, no traffic-related convictions or alcohol-influenced behavioural disturbances.
* 1 or 0 points on the modified Apfel scale for predicting post-operative nausea/vomiting (non-smoker, previously experienced nausea/vomiting post-operatively, previously experienced motion sickness)

Exclusion Criteria:

* Females (risk of teratogenicity)
* Non-caucasian ethnicity (possibility of deviant ethanol metabolism)
* Previous strong reactions such as nausea, fainting etc. during blood sampling
* Previous abnormal reactions to ethanol
* Previous convictions related to drug intoxication
* Previous excessive drug use
* Regular use of prescription drugs
* Two points or more according to the modified Apfel criteria

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Standard deviation of lateral position on road (SDLP) | Instantly (while the subject is inebriated)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Slørdal, PhD, MD, Principal Investigator — Norwegian University of Science and Technology; Gunnar D Jenssen, Principal Investigator — SINTEF Health Research
Locations (1):
- SINTEF Health and Research, Trondheim, Norway

REFERENCES:
- [Result] Helland A, Jenssen GD, Lervag LE, Westin AA, Moen T, Sakshaug K, Lydersen S, Morland J, Slordal L. Comparison of driving simulator performance with real driving after alcohol intake: a randomised, single blind, placebo-controlled, cross-over trial. Accid Anal Prev. 2013 Apr;53:9-16. doi: 10.1016/j.aap.2012.12.042. Epub 2013 Jan 28. PMID 23357031
- [Result] Helland A, Jenssen GD, Lervag LE, Moen T, Engen T, Lydersen S, Morland J, Slordal L. Evaluation of measures of impairment in real and simulated driving: Results from a randomized, placebo-controlled study. Traffic Inj Prev. 2016;17(3):245-50. doi: 10.1080/15389588.2015.1065975. Epub 2015 Jul 6. PMID 26147898